CLINICAL TRIAL: NCT00167934
Title: Metabolic Effects of Valproate and Antipsychotic Therapy
Brief Title: Determining Metabolic Effects of Valproate and Antipsychotic Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K23MH067795 (NIH); K23MH067795 (NIH); DAHBR AK-TNET1
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Results first posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-01

CONDITIONS: Schizophrenia
Keywords: Diabetes; Metabolic
MeSH Terms: conditions — Schizophrenia; Diabetes Mellitus | interventions — Valproic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): 50% of participants will receive placebo
  Interventions: Drug: Placebo
- Experimental (Experimental): 50% of participants will receive Depakote ER
  Interventions: Drug: Valproate

INTERVENTIONS:
Drug: Valproate — Depakote ER 500 mg to 3000 mg taken every night
  Other Names: Depakote ER
  Arms: Experimental
Drug: Placebo — Placebo given at same frequency as Valproate
  Arms: Placebo

SUMMARY:
This study will determine the metabolic processes responsible for high levels of blood glucose, metabolism disorders, and weight gain in people with schizophrenia who have been treated with antipsychotic medications in combination with valproate.

DETAILED DESCRIPTION:
This project aims to study the whole-body metabolic processes responsible for hyperglycemia, dyslipidemia and increased adiposity in schizophrenia patients treated with antipsychotic medications in combination with valproate. The project hypothesizes that combined treatment with valproate and antipsychotic medications will decrease insulin sensitivity at the level of skeletal muscle, liver and adipose tissue, in comparison to antipsychotic monotherapy. The decrease in insulin sensitivity is hypothesized to be associated with defects in glucose and lipid metabolism and increased adiposity

Treatment effects of antipsychotic/valproate combination therapy on different components of insulin secretion and action, and treatment effects on abdominal versus peripheral adiposity, are unknown despite the availability of gold-standard methods and the prognostic significance of these issues. Relevant data are needed to target basic research, to identify the potential for acute and long-term complications, and to plan therapeutic interventions. The following specific aims will be addressed in non-diabetic schizophrenia patients treated with atypical antipsychotics who will be randomized to open label treatment with either valproate or no adjuvant. Evaluations are performed at baseline and 3 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for schizophrenia, any type, treated with the same antipsychotic for at least 6 months
* No antipsychotic medication dose changes for 1 month, and no other medication changes for 1 month prior to study entry

Exclusion Criteria:

* Meets DSM-IV criteria for substance abuse within 3 months of study entry
* Involuntary legal status (as per Missouri law)
* Any serious medical disorder that may confound the assessment of relevant biologic measures or diagnosis, including: significant organ system dysfunction, metabolic diseases, type 1 or 2 diabetes mellitus, pregnancy, endocrine disease, coagulopathy, anemia, or acute infection
* Currently taking more than one antipsychotic medication
* Currently taking prescription medications (except certain psychotropic medications as discussed below), including oral contraceptive pills, any glucose lowering agent, lipid lowering agent, exogenous testosterone, recombinant human growth hormone, or any other endocrine agent that might confound substrate metabolism

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 164 (Actual)
Dates: Start 2004-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan W. Haupt, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Haupt DW, Newcomer JW. Hyperglycemia and antipsychotic medications. J Clin Psychiatry. 2001;62 Suppl 27:15-26; discussion 40-1. PMID 11806485
- See also: Click here for the Washington University Department of Psychiatry — http://www.psychiatry.wustl.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Experimental
Started | 82 | 82
Completed | 82 | 82
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline population consists of those participants who enrolled and completed the study. In other words, these are the participants that are included in the analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Experimental | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (10.1) | 41.3 (8.4) | 40.9 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 18 | 19 | 37
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 6 | 7 | 13
  African American | 19 | 18 | 37

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Body Fat Composition Using Dual Energy X-ray Absorptiometry at 12 Weeks
Description: Change in body composition (total body fat) was assessed using dual energy x-ray absorptiometry
Time Frame: Measured at baseline and Week 12
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Experimental
Number analyzed (Participants) | 24 | 22
percent change | -0.51 (2.13) | 2.03 (2.17)
Statistical Analysis 1: Comparison: Placebo vs Experimental; Test type: Superiority or Other; p < 0.0001, ANCOVA

2. Primary Outcome: Effects of Medication on Insulin Secretion at Skeletal Muscle (Glucose Disposal)
Time Frame: Measured at baseline and Week 12
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Experimental
Number analyzed (Participants) | 25 | 25
percent change | 0.27 (1.23) | -0.35 (1.13)
Statistical Analysis 1: Comparison: Placebo vs Experimental; Test type: Superiority or Other; p = 0.04, ANCOVA

ADVERSE EVENTS:
Time Frame: At 12 Week Assessment
Description: An Adverse Event Form is administered to participants by a trained rater.
Arm/Group | Placebo | Experimental
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 4/23 | 12/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=23) | Experimental (N=24)
Drowsiness/Somnolence (General disorders) | 1 | 2
Tiredness/Fatigue (General disorders) | 0 | 3
Anxiety (General disorders) | 1 | 2
Restlessness (General disorders) | 2 | 2
Tremor (General disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes